CLINICAL TRIAL: NCT00280111
Title: Reactogenicity and Immunogenicity of Live Attenuated Indian Rotavirus Vaccine Candidate Strains 116E and I321 in Healthy Non-Malnourished Infants 8-12 Weeks of Age
Brief Title: Safety and Immunogenicity Study of Live Attenuated Indian Rotavirus Vaccine Candidate Strains 116E and I321 in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: All India Institute of Medical Sciences (Other); National Institutes of Health (NIH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Stanford University (Other); Indian Institute of Science (Other Government); Children's Hospital Medical Center, Cincinnati (Other); Ministry of Science and Technology, India (Other Government); PATH (Other)
Responsible Party: Dr. MK Bhan, Dr. Pratima Ray, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 03-153; U01AI053719-02 (NIH)
Record Dates: First submitted 2006-01-13; First posted 2006-01-20 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: Rotavirus Infections
Keywords: rotavirus; vaccine; safety; immunogenicity; infants
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 116E AGMK
  Interventions: Biological: 116E AGMK
- 2 (Experimental): I321 AGMK
  Interventions: Drug: I321
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: 116E AGMK — Single dose of 116E 10^5 FFu
  Arms: 1
Drug: I321 — Single dose of I321 10^5 FFu
  Arms: 2
Drug: Placebo — 1 crystal of potassium permanganate dissolved in the bicarbonate buffer to colour match the vaccine
  Arms: 3

SUMMARY:
It has been observed that in children who get a severe rotavirus infection, subsequent infections cause either no symptoms or generally only mild or moderate diarrhea. This evidence is the basis for developing a vaccine since it suggests that the first infection immunizes the child against disease upon re-infection.

It was found that neonatal avirulent strains 116E and I321 induce protective immunity and offer clinical protection for at least one year. Both these strains are well characterized and the safety studies have been done in animal models. These candidate vaccine strains have been evaluated for safety and immunogenicity in adults and children (2 to 12 years of age) by a randomized double blind placebo controlled trial in Cincinnati, USA. In India, the diversity of rotavirus strains is greater and there is greater prevalence of malnutrition and co-infection with other enteric pathogens. These vaccines have therefore, also been tested in India.

DETAILED DESCRIPTION:
This study was a phase I randomized, double blind, safety and immunogenicity study of live, attenuated neonatal rotavirus vaccine candidate strains 116E or I321 in healthy non-malnourished infants aged 8-12 weeks. Informed, written, witnessed consent was obtained from the parents before infants were screened at 6 weeks of age. Infants (n=90) were randomized (30 per group) to receive one dose of either the 116E or I321 vaccines (10^5 fluorescence focus units, FFu) or placebo at 8 weeks of age. The rotavirus vaccine was administered at a different time than DPT (Diptheria-Pertussis-Tetanus), OPV (Oral Polio Vaccine) and HBV (Hepatitis B vaccine) immunization since the trial represented the first safety study in infants with these strains. The DPT, OPV and HBV vaccines were given at the regular EPI schedule of 6, 10 and 14 weeks with the precautions and techniques routinely in place for these.

The test article was administered orally two weeks after the first DPT, OPV and HBV dose, after half an hour of administering 2.5 ml bicarbonate to buffer stomach acidity.

Evaluation of reactogenicity consisted of daily recording of symptoms reported by the mother/caregiver and twice-daily axillary temperature measurements for 14 days post administration of vaccine/placebo. Stool specimens were collected before administration of vaccine/placebo, twice during the week following administration (days 3 and 7), and at day 28 after administration to evaluate for vaccine virus shedding. Weekly recording of adverse events was also done for the next 2 weeks i.e. on days 21 and 28 post administration of vaccine/placebo. If gastrointestinal signs or symptoms occurred any time during the 4 weeks observation period, attempts were made to collect stool samples daily (maximum 2 per day) while the illness persisted, to be examined for the presence of the vaccine strains.

Immunogenicity was determined by analysis of sera obtained before immunization and 28 days after immunization for changes in titers of rotavirus antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants
* Consent available

Exclusion Criteria:

* Evidence of renal, cardiovascular, liver or other reticuloendothelial, neurological, gastrointestinal, hematologic, rheumatologic or immunologic disease

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
- Safety | 4 weeks after test article administration

SECONDARY OUTCOMES:
- Vaccine Take, antibody titers in subjects in vaccine and placebo groups 28 days after administration of vaccine/placebo or shedding of rotavirus vaccine strains by antigen detection ELISA on days 3, 7 and 28 post administration. | 4 weeks post administration of test article

CONTACTS AND LOCATIONS:
Overall Officials: Maharaj K Bhan, MD, Principal Investigator — All India Institute of Medical Sciences; Pratima Ray, PhD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Society for Applied Studies, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Bhandari N, Sharma P, Glass RI, Ray P, Greenberg H, Taneja S, Saksena M, Rao CD, Gentsch JR, Parashar U, Maldonado Y, Ward RL, Bhan MK. Safety and immunogenicity of two live attenuated human rotavirus vaccine candidates, 116E and I321, in infants: results of a randomised controlled trial. Vaccine. 2006 Jul 26;24(31-32):5817-23. doi: 10.1016/j.vaccine.2006.05.001. Epub 2006 May 12. PMID 16735085